CLINICAL TRIAL: NCT00375180
Title: Nutritional Status and Barriers to Dietary Intake in Head and Neck Cancer Patients Prior to, on Completion of and Six Weeks After Oncology Treatment
Brief Title: Nutritional Status and Barriers to Dietary Intake in Head and Neck Cancer Patients
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HN-4-0030 / 23028
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-03

CONDITIONS: Head and Neck Cancer
Keywords: food; diet; mucositis; xerostomia; dysphagia; taste; smell; head and neck; radiation; chemotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis; Xerostomia; Deglutition Disorders; Anosmia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators hope to learn more about how side-effects of RT or RTchemo affect food intake and nutrition status.

DETAILED DESCRIPTION:
Head and neck cancer patients often have difficulty meeting their nutritional needs while undergoing radiation therapy (RT) and/or chemotherapy (RTchemo). Tumor locations and side effects of RT or RTchemo, including dry mouth, mouth sores, difficulty chewing and swallowing, changes in taste and smell, and loss of appetite, lead to poor food intake and weight loss. The investigators hope to learn more about how side-effects of RT or RTchemo affect food intake and nutrition status.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosed with head and neck cancer including the lip, oral cavity, salivary glands, paranasal sinuses, oropharynx, nasopharynx, hypopharynx, larynx, and thyroid
* All histological types of cancer
* All tumour stages according to American Joint Committee for Cancer (AJCC) Staging
* All forms of RT including standard or investigational and/or concurrent standard or investigational chemotherapy for head and neck cancers
* Alert and mentally competent
* English speaking

Exclusion Criteria:

* Unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed with head and neck cancer including the lip, oral cavity, salivary glands, paranasal sinuses, oropharynx, nasopharynx, hypopharynx, larynx, and thyroid
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vickie Baracos, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada